CLINICAL TRIAL: NCT05089058
Title: Lóa Project: An Exploratory Pilot Randomised Controlled Trial of a Remotely-delivered Brief Cognitive Intervention to Reduce Intrusive Memories of Trauma for Women in Iceland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Andri Steinþór Björnsson, Professor, University of Iceland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-214
Record Dates: First submitted 2021-10-05; First posted 2021-10-22 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Intrusive Memories of Traumatic Event(s)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief cognitive task (delivered digitally) (Experimental)
  Interventions: Behavioral: Brief, digitally delivered imagery-competing task intervention package, comprised of:
- Brief relaxation exercise task (delivered digitally) (Placebo Comparator)
  Interventions: Behavioral: Brief, digitally delivered relaxation task intervention, comprised of:

INTERVENTIONS:
Behavioral: Brief, digitally delivered imagery-competing task intervention package, comprised of: — Two sessions guided (remotely) by a researcher. Sessions comprised of:
  (i) task procedure: a memory cue followed by playing imagery-competing computer game task with mental rotation instructions. Monitoring of intrusive memories to select hotspot cue, and which intrusion to target.
  (ii) accompanying information, including rationale for the brief cognitive task.
  (iii) option to use the brief cognitive task after the session (self-administered); option to engage in up to 6 guided booster sessions supported by a researcher.
  Arms: Brief cognitive task (delivered digitally)
Behavioral: Brief, digitally delivered relaxation task intervention, comprised of: — Brief, digitally delivered relaxation task intervention, comprised of:
  Two sessions guided (remotely) by a researcher. Sessions comprised of:
  (i) relaxation exercise task using instruction components from progressive muscle relaxation
  (ii) accompanying information, including rationale for the brief relaxation exercise task.
  (iii) option to use the brief relaxation exercise task after the session (self-administered); option to engage in up to 6 guided booster sessions supported by a researcher.
  Arms: Brief relaxation exercise task (delivered digitally)

SUMMARY:
Intrusive memories are sensory memories of a traumatic event(s) that spring to mind involuntarily, evoke strong emotions, and disrupt functioning in daily life. Previous research has demonstrated that a brief cognitive intervention can prevent the development of intrusive memories as well as reduce the number of intrusive memories of long-standing trauma. Initial pilot work (using case studies) with women in Iceland indicates that the intervention is acceptable and feasible.

This exploratory pilot trial will compare remote delivery of the intervention (i.e. brief, digitally delivered imagery-competing task intervention, n = 12) to an attention-placebo control condition (i.e., brief, digitally delivered relaxation exercise task; n = 12). We will explore whether (relative to the control condition) the intervention: (i) reduces the number of intrusive memories (primary outcome), and (ii) improves other symptoms and functioning.

This study is funded by the OAK foundation (OCAY-18-442) and the Strategic Research and Development Program: Societal Challenges in Iceland (200095-5601).

DETAILED DESCRIPTION:
The proposed study will involve a brief intervention (c. 2 guided sessions with the researcher; options for up to 6 additional booster sessions) delivered digitally and remotely (i.e., not physically in-person), and with initial guided support (remotely delivered) from a researcher. Participants will be asked to fill out a diary indicating the number of intrusive memories they experienced, along with self-report questionnaires, at baseline (i.e., one week prior to commencement of the intervention), week 1 (week after the second intervention/control session), week 5 (primary outcome; 5 weeks from the second intervention/control session), and at 1-, 3- and 6-months follow-up.

Monitoring will be performed by a clinical trial unit to verify that the study is conducted and data are generated and documented in compliance with GCP and the applicable regulatory requirements.

Potentially eligible participants for this pilot study will be identified using data collected in the SAGA cohort study (an epidemiological study of trauma among Icelandic women).

ELIGIBILITY:
Inclusion Criteria:

* Aged: 18-69 (at time of enrollment to cohort study)
* Able to speak and read study materials in Icelandic or English
* Willing to be contacted remotely and having access to a smartphone or computer
* Experienced intrusive memories in past month (PCL-5 item 1 score is ≥ 2)
* Experienced 2 or more intrusive memories of a traumatic event in the past week
* Willing to monitor intrusive memories in everyday life
* Willing and able to complete remote study sessions

Exclusion Criteria:

* Suicide risk indicated in the initial assessment (response of 'nearly every day' to item 9 on PHQ-9) and by responses on MINI during follow-up telephone risk assessment

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories of traumatic event(s) | Week 5
  Number of intrusive memories of traumatic event(s) recorded in a brief daily diary for 7 days

SECONDARY OUTCOMES:
Number of intrusive memories of traumatic event(s) | Baseline, Week 1, Week 12 and Week 24
  Number of intrusive memories of traumatic event(s) recorded in a brief daily diary for 7 days
The Posttraumatic Stress Disorder Checklist 5 (PCL-5) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  A 20-item questionnaire assessing the severity of PTSD symptoms corresponding to the DSM-5 criteria for PTSD. Symptoms are rated on a 5-point Likert-scale.
The Patient Health Questionnaire-9 (PHQ-9) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  A 9-item questionnaire assessing depression symptoms and their severity. Items are scored from 0 (i.e., not at all) to 3 (i.e., nearly every day).
The Generalized Anxiety Disorder-7 scale (GAD-7) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  A 7-item questionnaire designed as a screening tool for symptoms of GAD and their severity. Items are scored from 0 (i.e., not at all) to 3 (i.e., nearly every day).
Characteristics of intrusive memories | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  6 self-rated items assessing the frequency of unwanted memories of the trauma in the previous week (on a 7-point scale, from never to many times a day) and the level of distress, nowness, reliving, disconnectedness and whether different triggers are associated with unwanted trauma memories (on an 11-point scale, from 0 to 100). Higher scores indicate more unwanted memories, higher levels of distress/nowness/reliving/disconnectedness and more different triggers.
Impact of intrusive memories on concentration, sleep and stress | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  Assessed with six self-rated items anchored to the past week: two items assessing concentration difficulties in general and due to intrusive memories (11-point scale; high scores indicating more difficulties), one item assessing duration of disruption after experiencing intrusive memory (<1 minute to > 60 minutes), two items assessing sleep disturbance due to intrusive memories (11-point scale; higher scores indicating more sleep disturbance) and one item assessing the degree to which intrusive memories affected stress levels (0 = not at all; 10 = very much).
General impact of intrusive memories | Baseline, Week 1, Week, 5, Week 12 and Week 24
  Assessed with two self-rated items, one assessing the degree of distress associated with intrusive memories and the other assessing how vivid they were in the past week (both rated on an 11-point scale, 0 = not at all; 10 = very distressing; 0 = not at all; 10 = very vivid).
Impact of intrusive memories on daily functioning | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  Assessed with four items. One question is self-rated: "Have the intrusive memories affected your ability to function in your daily life?" on an 11-point scale; higher score indicating greater impact on functioning. The other question is open-ended: "How have the intrusive memories affected your ability to function in your daily life in the past week?"). We will also explore whether there is a link between the content of participants' intrusive memories and specific domains of functioning - in open-ended discussion and using questions (asked at baseline) such as: "Are there any specific activities that you would like to do, but avoid because they are linked to your intrusive memories?" and "What change in your intrusive memories would make a meaningful difference in your life?" along with (asked at follow-ups, after the intervention/control task) "Since starting the study, are there any specific activities that you used to avoid (due to your intrusive memories), but now do more often?"
The Sheehan Disability Scale (SDS) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  A self-report questionnaire assessing functional impairment across three domains: (1) Work/school, (2) social, and (3) family life. Domains are measured on an 11-point Likert scale, ranging from 0 (i.e., not at all) to 10 (i.e., extremely). The scale will be adapted to assess functional impairment associated with intrusive memories.
The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  A 12-item questionnaire assessing difficulties due to health conditions, including mental or emotional problems (with reference to study event). Scores range from 1 ("none") to 5 ("extremely/cannot do"). Lower scores indicate better functioning.
The Psychological Outcome Profiles; PSYCHLOPS | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  A 4-item a patient-generated outcome measure of symptom-change after therapy/interventions, consisting of four items measuring three domains: problems (two items), function (one item), and well-being (one item). The patient chooses which symptoms or problems are most important to measure over the course of an intervention.
Self-rated Health rating (SRHR) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  A single item assessing perceived health status on a 4-point scale (very good to very bad). The scale is reverse-scored; higher scores indicate better health.
The Pittsburgh Sleep Quality Index Addendum for PTSD (PSQI-A) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  A 7-item self-report questionnaire assessing the frequency of disruptive nocturnal behaviours (e.g., acting out dreams, episodes of terror or screaming) common in PTSD. Respondents report symptoms over the past month on a 4-point Likert scale, ranging from 0 (never in the past month) to 3 (three or more times each week). Total score ranges from 0 to 21. A clinical score ≥ 4 will be used, which discriminates between participants with and without PTSD.
Sleep Condition Indicator (SCI-2) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  2 self-rated items; one assesses the extent to which the respondent is experiencing poor sleep (with reference to study event) on a 5-point scale (from not at all to very much), one assesses the number of nights in the week the respondent experiences sleep problems on 5-point scale (from 0-1 to 5-7 nights). Both 5-point scales are reverse scored (0 - 4) then summed. Possible total scores range from 0-8; higher values indicate better sleep.
Time Perspective Questionnaire (TPQ) | Baseline, Week 1, and 1-month, 3-month and 6-month follow-ups
  8-items drawn or modified from both the Temporal Orientation Scale and the Zimbardo Time Perspective Inventory. Respondents rate how true statements are for them on a 5-point scale, from not at all true (1) to very true (5) (e.g., "My plans about the future are pretty well laid out", "It is best to live day-to-day").

OTHER OUTCOMES:
Credibility/expectancy scale. | First intervention session = 7 days from baseline, Week 1 and Week 5
  Prior to completing the intervention, participants provide 4 ratings of treatment expectancy and the degree to which they found the intervention credible in both conditions.
Vividness of visual imagery question (adapted from VVIQ-2) | First intervention session = 7 days from baseline
  A self-rated item assessing the degree of vividness/clarity of a trauma memory after it is brought to mind during the first part of the intervention. Responses are scored on a 5-point scale from 1=no image at all to 5=perfectly clear and vivid as normal vision). In intervention arm only.
Acceptability and feasibility | Week 1, 1-month, and 3-month follow-ups
  Self-rated questions assessing acceptability and feasibility of the intervention/control tasks (e.g., ratings of the extent to which the respondent would recommend the intervention, whether they consider it to be an acceptable way to reduce the frequency of intrusive memories). We will also include two self-rated and one open-ended question about the experience of using the digital platform to complete study procedures.
Intrusion diary adherence | Week 1, Week 5, Week 12 and Week 24
  A self-rated item assessing self-reported accuracy of filling out the diary (0 = not at all; 10 = very accurately).
Adverse Events (AEs). | Week 1, and 1-month, 3-month and 6-month follow-ups
  Participants will be asked whether they had experienced any adverse events with one open-ended question: 'Have you had any health problems since the last contact?'

CONTACTS AND LOCATIONS:
Overall Officials: Andri Björnsson, Principal Investigator — University of Iceland; Emily Holmes, Principal Investigator — Uppsala University
Locations (1):
- University of Iceland, Sæmundargata 12, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Anonymised research data will be made available on Open Science Framework (OSF) indefinitely.
  OSF is an open source web application that is freely accessible to public and scientific community.